CLINICAL TRIAL: NCT03686007
Title: A Multimedia Self-management Intervention to Prepare Family Caregivers and Patients for Lung Cancer Surgery
Brief Title: Multimedia Self-Management Intervention for Lung Cancer Surgery Family Caregivers and Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17238; NCI-2017-01391 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 17238 (Other: City of Hope Medical Center)
Record Dates: First submitted 2017-08-01; First posted 2018-09-26 (Actual); Results first posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Caregiver; Stage I Lung Cancer AJCC v7; Stage IA Lung Cancer AJCC v7; Stage IB Lung Cancer AJCC v7; Stage II Lung Cancer AJCC v7; Stage IIA Lung Cancer AJCC v7; Stage IIB Lung Cancer AJCC v7; Stage III Lung Cancer AJCC v7; Stage IIIA Lung Cancer AJCC v7; Stage IIIB Lung Cancer AJCC v7
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (MSM intervention) (Experimental): Patients and FCGs receive the MSM intervention consisting of videos, a handbook, and research nurse coaching over 40-60 minutes, approximately 3-7 days before surgery and within 24 hours of planned discharge. Patients and FCGs also receive research nurse support via telephone(separate sessions for FCGs and patients) over 20-30 minutes at 2 and 7 days, and 2 months post-discharge.
  Interventions: Other: Informational Intervention; Other: Media Intervention
- Group II (Attention Control) (Active Comparator): Patients and FCGs receive attention control intervention consisting of videos (American Cancer Society video on "Clinical Trials"), American Cancer Society print materials, and assistance from a CRA approximately 3-7 days before surgery and within 24 hours of planned discharge. Patients and FCGs also receive assistance from CRAs via telephone at 2 and 7 days, and 2 months post-discharge.
  Interventions: Other: Informational Intervention; Other: Media Intervention

INTERVENTIONS:
Other: Informational Intervention — Receive MSM intervention handbook
  Arms: Group I (MSM intervention)
Other: Informational Intervention — Receive MSM intervention research nurse coaching
  Arms: Group I (MSM intervention)
Other: Informational Intervention — Receive ASCO print materials
  Arms: Group II (Attention Control)
Other: Informational Intervention — Receive CRA assistance
  Arms: Group II (Attention Control)
Other: Media Intervention — View the MSM intervention videos
  Arms: Group I (MSM intervention)
Other: Media Intervention — View American Cancer Society (ACS) videos
  Arms: Group II (Attention Control)

SUMMARY:
This randomized phase III trial studies how well a multimedia self-management intervention works in preparing family caregivers and patients with stage I-III lung cancer for lung cancer surgery. The multimedia self-management intervention, Preparing for your Lung Cancer Surgery, is a nurse-led, caregiver-based, multimedia intervention that may improve patient recovery after surgery, lower caregiving burden, and improve distress and quality of life.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Test the effects of the multimedia self-management (MSM) intervention on family caregivers (FCG) outcomes and cancer support services use at discharge and 3-month post-discharge, comparing intervention and attention control groups.

II. Test the effects of the MSM intervention on patient outcomes and healthcare resource use at discharge and 3-months post-discharge, comparing intervention and attention control groups.

III. Test the effects of the MSM intervention on outcome mediators at discharge and 3-months post-discharge, comparing intervention and attention control groups.

SECONDARY OBJECTIVES:

I. Explore moderators (age, sex, marital status, caregiver relationship to patient, caregiver employment status, co-morbidities) of FCG and patient outcomes and reciprocal relationships.

II. Determine, through exit interviews, participant's experience with the MSM intervention.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients and FCGs receive the MSM intervention consisting of videos, a handbook, and research nurse coaching over 40-60 minutes, approximately 3-7 days before surgery and within 24 hours of planned discharge. Patients and FCGs also receive research nurse support by telephone (separate sessions for FCGs and patients) over 20-30 minutes at 2 and 7 days, and 2 months post-discharge.

GROUP II: Patients and FCGs receive attention control intervention consisting of videos (American Cancer Society video on "Clinical Trials"), American Cancer Society print materials, and assistance from a clinical research associate (CRA) approximately 3-7 days before surgery and within 24 hours of planned discharge. Patients and FCGs also receive assistance from CRAs via telephone calls at 2 and 7 days, and 2 months post-discharge.

ELIGIBILITY:
Family Caregiver Inclusion Criteria:

* A family member or friend identified by the patient as being the primary care provider before and after surgery
* A patient/care recipient enrolled in the study
* Age 21 years or older
* Able to read or understand English

Patient Inclusion Criteria:

* Diagnosis of Stage I-III non-small cell lung cancer
* Scheduled to undergo surgery for treatment
* A family caregiver enrolled in the study
* Age 21 years or older
* Able to read or understand English.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2018-11-06 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2026-01-13 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Sun, RN, PhD, Principal Investigator — City of Hope Medical Center; Jae Kim, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

REFERENCES:
- [Derived] Sun V, Raz DJ, Erhunmwunsee L, Ruel N, Carranza J, Prieto R, Ferrell B, Krouse RS, McCorkle R, Kim JY. Improving family caregiver and patient outcomes in lung cancer surgery: Study protocol for a randomized trial of the multimedia self-management (MSM) intervention. Contemp Clin Trials. 2019 Aug;83:88-96. doi: 10.1016/j.cct.2019.07.002. Epub 2019 Jul 3. PMID 31279090

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 542 participants (342 patients, 200 caregivers) were assessed for study eligibility. After 162 participants were excluded for various reasons - not meeting inclusion criteria (n= 91), declined to participate (n= 48), other/unknown reasons (n= 3), late ineligibility (n= 20), 380 participants (190 dyads - 190 patients, 190 caregivers) were randomized.
Pre-assignment Details: 542 participants (342 patients, 200 caregivers) were assessed for study eligibility. After 162 participants were excluded for various reasons - not meeting inclusion criteria (n= 91), declined to participate (n= 48), other/unknown reasons (n= 3), late ineligibility (n= 20), 380 participants (190 dyads - 190 patients, 190 caregivers) were randomized.
Groups:
- Group I (MSM Intervention): Patients and FCGs receive the MSM intervention consisting of videos, a handbook, and research nurse coaching over 40-60 minutes, approximately 3-7 days before surgery and within 24 hours of planned discharge. Patients and FCGs also receive research nurse support via telephone(separate sessions for FCGs and patients) over 20-30 minutes at 2 and 7 days, and 2 months post-discharge.
  Informational Intervention: Receive MSM intervention handbook
  Informational Intervention: Receive MSM intervention research nurse coaching
  Media Intervention: View the MSM intervention videos
  Quality-of-Life Assessment: Ancillary studies
  Questionnaire Administration: Ancillary studies
- Group II (Attention Control): Patients and FCGs receive attention control intervention consisting of videos (American Cancer Society video on "Clinical Trials"), American Cancer Society print materials, and assistance from a CRA approximately 3-7 days before surgery and within 24 hours of planned discharge. Patients and FCGs also receive assistance from CRAs via telephone at 2 and 7 days, and 2 months post-discharge.
  Informational Intervention: Receive ASCO print materials
  Informational Intervention: Receive CRA assistance
  Media Intervention: View ASCO Cancer.net videos
Period: Overall Study
Arm/Group | Group I (MSM Intervention) | Group II (Attention Control)
Started | 188 (94 dyads, consisting of 94 patients and 94 caregivers were randomized to the intervention arm.) | 192 (96 dyads, consisting of 96 patients and 96 caregivers were randomized to the control arm.)
Completed | 156 (82 dyads, consisting of 81 patients and 75 caregivers completed follow-up. This number (82 dyads) includes incomplete dyads e.g. cases where the patient completed follow-up and the caregiver was lost to follow-up.) | 155 (80 dyads, consisting of 79 patients and 76 caregivers completed follow-up. This number (80 dyads) includes incomplete dyads e.g. cases where the patient completed follow-up and the caregiver was lost to follow-up.)
Not Completed | 32 | 37

BASELINE CHARACTERISTICS:
Population: This baseline table includes data for patients and caregivers.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group I (MSM Intervention) | Group II (Attention Control) | Total
Number analyzed (Participants) | 188 | 192 | 380
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 67.5 [60.0 to 74.0] | 65.0 [53.0 to 74.0] | 66.0 [56.0 to 74.0]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Due to missing item responses and no separate category for "Unknown" sex, the number of participants analyzed differs from the overall number of participants.
  Participants
    number analyzed (Participants) | 187 | 192 | 379
    Female | 110 | 116 | 226
    Male | 77 | 76 | 153
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27 | 21 | 48
  Not Hispanic or Latino | 153 | 166 | 319
  Unknown or Not Reported | 8 | 5 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 42 | 43 | 85
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 4 | 8 | 12
  White | 126 | 118 | 244
  More than one race | 1 | 6 | 7
  Unknown or Not Reported | 13 | 16 | 29
Region of Enrollment [Number; unit: participants]
  United States | 188 | 192 | 380

OUTCOME MEASURES:

1. Primary Outcome: Change in Family Caregiver Psychological Distress (as Measured by the Distress Thermometer)
Description: Mean caregiver psychological distress scores from baseline to 3 months post-discharge were calculated. A linear mixed-effects model was used to assess differences in psychological distress between the intervention and control arm over time.
  Score range: 0-10. Higher score means worse outcome.
Time Frame: Outcomes are measured at baseline, 1 month, and 3 months post-discharge. Absolute values are reported at each timeframe.
Population: Due to attrition in the study, the number of family caregivers assessed at baseline differs from the number of family caregivers analyzed during follow-up.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Group I (MSM Intervention) | Group II (Attention Control)
Number analyzed (Participants) | 92 | 96
score on a scale
  Baseline | 3.92 [3.38 to 4.47] | 4.19 [3.65 to 4.72]
  1 month post-discharge: number analyzed (Participants) | 75 | 68
  1 month post-discharge | 3.38 [2.79 to 3.98] | 3.74 [3.12 to 4.36]
  3 months post-discharge: number analyzed (Participants) | 75 | 74
  3 months post-discharge | 3.22 [2.62 to 3.82] | 4.14 [3.54 to 4.74]

2. Primary Outcome: Change in Caregiving Burden (as Measured by the Montgomery Borgatta Caregiver Burden Scale)
Description: Mean caregiver burden scores from baseline to 3 months post-discharge were calculated. A linear mixed-effects model was used to assess differences in burden between the intervention and control arm over time. The model included treatment arm, time, and the interaction between treatment arm and time as effects.
  Total burden score is calculated by summing items from 3 subscales: objective burden, subjective burden & demand burden.
  Score range: 14-70. Higher score means worse outcome.
Time Frame: Outcomes are measured at baseline, 1 month, and 3 months post-discharge. Absolute values are reported at each timeframe.
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Group I (MSM Intervention) | Group II (Attention Control)
Number analyzed (Participants) | 93 | 95
score on a scale
  Baseline | 44.68 [43.01 to 46.35] | 44.56 [42.91 to 46.21]
  1 month post-discharge: number analyzed (Participants) | 75 | 68
  1 month post-discharge | 42.19 [40.36 to 44.02] | 44.73 [42.83 to 46.63]
  3 months post-discharge: number analyzed (Participants) | 76 | 76
  3 months post-discharge | 40.45 [38.63 to 42.27] | 42.00 [40.18 to 43.82]

3. Primary Outcome: Change in Preparedness for Caregiving (as Measured by the Preparedness for Caregiving Scale)
Description: Mean caregiver preparedness scores from baseline to 3 months post-discharge were calculated. A linear mixed-effects model was used to assess differences in preparedness between the intervention and control arm over time.
  Score range: 0-4. Higher score means better outcome.
Time Frame: Outcomes are measured before surgery (baseline), 1 month, and 3 months post-discharge. Absolute values are reported at each timeframe.
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Group I (MSM Intervention) | Group II (Attention Control)
Number analyzed (Participants) | 93 | 95
score on a scale
  Baseline | 2.55 [2.38 to 2.72] | 2.60 [2.44 to 2.77]
  1 month post-discharge: number analyzed (Participants) | 75 | 68
  1 month post-discharge | 2.98 [2.80 to 3.16] | 2.88 [2.70 to 3.07]
  3 months post-discharge: number analyzed (Participants) | 75 | 76
  3 months post-discharge | 2.94 [2.76 to 3.12] | 2.78 [2.60 to 2.96]

4. Primary Outcome: Change in Family Caregiver Quality of Life (as Measured by the City of Hope-Quality of Life-Family (COH-QOL-Family)
Description: Mean caregiver QoL scores from baseline to 3 months post-discharge were calculated. A linear mixed-effects model was used to assess differences in QoL between the intervention and control arm over time.
  Total QoL score is calculated by summing items from 3 subscales: physical well-being, psychological well-being, social concerns & spiritual well-being.
  Score range: 0-40. Higher score means better outcome.
Time Frame: Outcomes are measured at baseline, 1 month, and 3 months post-discharge. Absolute values are reported at each timeframe.
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Group I (MSM Intervention) | Group II (Attention Control)
Number analyzed (Participants) | 93 | 94
score on a scale
  Baseline | 27.04 [25.85 to 28.22] | 26.83 [25.65 to 28.01]
  1 month post-discharge: number analyzed (Participants) | 75 | 67
  1 month post-discharge | 27.69 [26.45 to 28.94] | 26.67 [25.40 to 27.94]
  3 months post-discharge: number analyzed (Participants) | 75 | 76
  3 months post-discharge | 27.51 [26.27 to 28.76] | 26.43 [25.20 to 27.67]

5. Primary Outcome: Number of Participants Who Used Family Caregiver Resource (as Measured by the Family Caregiver Healthcare Use Inventory)
Description: Differences in the number of caregivers who saw a support services specialist were compared between both groups using Chi-squared and Fisher's exact test.
Time Frame: Outcomes are measured at discharge, 1 month, and 3 months post-discharge.
Population: Due to attrition in the study, the number of family caregivers assessed at discharge differs from the number of family caregivers analyzed during follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (MSM Intervention) | Group II (Attention Control)
Number analyzed (Participants) | 90 | 94
Participants
  Discharge: number analyzed (Participants) | 88 | 94
  Discharge | 8 | 5
  1 month post-discharge: number analyzed (Participants) | 90 | 89
  1 month post-discharge | 2 | 0
  3 months post-discharge: number analyzed (Participants) | 89 | 93
  3 months post-discharge | 0 | 2

6. Primary Outcome: Change in Patient Psychological Distress (as Measured by the Distress Thermometer)
Description: Mean patient psychological distress scores from baseline to 3 months post-discharge were calculated. A linear mixed-effects model was used to assess differences in psychological distress between the intervention and control arm over time.
  Score range: 0-10. Higher score means worse outcome.
Time Frame: Outcomes are measured at baseline, 1 month, and 3 months post-discharge. Absolute values are reported at each timeframe.
Population: Due to attrition in the study, the number of patients assessed at baseline differs from the number of patients analyzed during follow-up.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Group I (MSM Intervention) | Group II (Attention Control)
Number analyzed (Participants) | 94 | 96
score on a scale
  Baseline | 4.23 [3.60 to 4.80] | 4.39 [3.80 to 5.00]
  1 month post-discharge: number analyzed (Participants) | 75 | 69
  1 month post-discharge | 3.42 [2.80 to 4.10] | 3.55 [2.90 to 4.20]
  3 months post-discharge: number analyzed (Participants) | 79 | 77
  3 months post-discharge | 3.25 [2.60 to 3.90] | 3.76 [3.10 to 4.40]

7. Primary Outcome: Change in Patient Quality of Life (as Measured by the Functional Assessment of Cancer Therapy-Lung - FACT-L)
Description: Mean patient QoL scores from baseline to 3 months post-discharge were calculated. A linear mixed-effects model was used to assess differences in QoL between the intervention and control arm over time.
  Total FACT-L score is calculated by summing items from 5 subscales: physical well-being, social/family well-being, emotional well-being, functional well-being & lung cancer subscale.
  Score range: 0-136. Higher score means better outcome.
Time Frame: Outcomes are measured at baseline, 1 month, and 3 months post-discharge. Absolute values are reported at each timeframe.
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Group I (MSM Intervention) | Group II (Attention Control)
Number analyzed (Participants) | 93 | 94
score on a scale
  Baseline | 106.09 [102.20 to 109.90] | 104.27 [100.40 to 108.10]
  1 month post-discharge: number analyzed (Participants) | 76 | 68
  1 month post-discharge | 103.97 [99.80 to 108.10] | 99.17 [94.90 to 103.50]
  3 months post-discharge: number analyzed (Participants) | 79 | 77
  3 months post-discharge | 103.54 [99.50 to 107.60] | 101.04 [96.90 to 105.20]

8. Primary Outcome: Number of Participants Who Used Patient Healthcare Resource Use (Home Health Nursing Care, Urgent/ER Visits, Hospital Readmissions)
Description: Differences in the number of patients who were readmitted to the hospital for an overnight stay were compared between both groups using Chi-squared and Fisher's exact test.
Time Frame: Outcomes are measured at 1 month, and 3 months post-discharge.
Population: Due to attrition in the study, the number of patients assessed differed during follow-up timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (MSM Intervention) | Group II (Attention Control)
Number analyzed (Participants) | 90 | 90
Participants
  1 month post-discharge | 4 | 2
  3 months post-discharge: number analyzed (Participants) | 81 | 78
  3 months post-discharge | 7 | 8

9. Secondary Outcome: Change in Family Caregiver Self-efficacy (as Measured by the Self-Efficacy Scale)
Description: Mean caregiver self-efficacy scores from baseline to 3 months post-discharge were calculated. A linear mixed-effects model was used to assess differences in self-efficacy between the intervention and control arm over time.
  Score range: 1-4. Higher score means better outcome.
Time Frame: Outcomes are measured at baseline, 1 month, and 3 months post-discharge. Absolute values are reported at each timeframe.
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Group I (MSM Intervention) | Group II (Attention Control)
Number analyzed (Participants) | 92 | 93
score on a scale
  Baseline | 3.33 [3.22 to 3.44] | 3.33 [3.22 to 3.44]
  1 month post-discharge: number analyzed (Participants) | 74 | 67
  1 month post-discharge | 3.47 [3.35 to 3.59] | 3.38 [3.25 to 3.50]
  3 months post-discharge: number analyzed (Participants) | 74 | 75
  3 months post-discharge | 3.52 [3.41 to 3.64] | 3.40 [3.28 to 3.52]

10. Secondary Outcome: Change in Patient Self-efficacy (as Measured by the Self-Efficacy Scale)
Description: Mean patient self-efficacy scores from baseline to 3 months post-discharge were calculated. A linear mixed-effects model was used to assess differences in self-efficacy between the intervention and control arm over time.
  Score range: 1-4. Higher score means better outcome.
Time Frame: Outcomes are measured at baseline, 1 month, and 3 months post-discharge. Absolute values are reported at each timeframe.
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Group I (MSM Intervention) | Group II (Attention Control)
Number analyzed (Participants) | 94 | 94
score on a scale
  Baseline | 3.60 [3.50 to 3.70] | 3.51 [3.40 to 3.60]
  1 month post-discharge: number analyzed (Participants) | 76 | 69
  1 month post-discharge | 3.60 [3.50 to 3.70] | 3.52 [3.40 to 3.60]
  3 months post-discharge: number analyzed (Participants) | 78 | 76
  3 months post-discharge | 3.56 [3.50 to 3.70] | 3.55 [3.40 to 3.70]

11. Secondary Outcome: Change in Family Caregiver Activation (as Measured by the FCG Activation in Transitions Tool)
Description: Mean caregiver activation scores from baseline to 3 months post-discharge were calculated. A linear mixed-effects model was used to assess differences in activation between the intervention and control arm over time.
  Score range: 10-60. Higher score means better outcome.
Time Frame: Outcomes are measured at baseline, 1 month, and 3 months post-discharge. Absolute values are reported at each timeframe.
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Group I (MSM Intervention) | Group II (Attention Control)
Number analyzed (Participants) | 93 | 93
score on a scale
  Baseline | 46.33 [44.30 to 48.37] | 47.30 [45.27 to 49.33]
  1 month post-discharge: number analyzed (Participants) | 75 | 67
  1 month post-discharge | 48.50 [46.34 to 50.67] | 48.76 [46.54 to 50.99]
  3 months post-discharge: number analyzed (Participants) | 75 | 76
  3 months post-discharge | 47.79 [45.62 to 49.96] | 48.37 [46.22 to 50.53]

12. Secondary Outcome: Change in Patient Activation (as Measured by the Patient Activation Measure)
Description: Mean patient activation scores from baseline to 3 months post-discharge were calculated. A linear mixed-effects model was used to assess differences in activation between the intervention and control arm over time.
  Score range: 0-100. Higher score means better outcome.
Time Frame: Outcomes are measured at baseline, 1 month, and 3 months post-discharge. Absolute values are reported at each timeframe.
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Group I (MSM Intervention) | Group II (Attention Control)
Number analyzed (Participants) | 94 | 95
score on a scale
  Baseline | 73.30 [69.70 to 76.90] | 71.51 [67.90 to 75.10]
  1 month post-discharge: number analyzed (Participants) | 77 | 69
  1 month post-discharge | 75.41 [71.60 to 79.30] | 71.00 [67.00 to 75.00]
  3 months post-discharge: number analyzed (Participants) | 80 | 76
  3 months post-discharge | 74.47 [70.70 to 78.30] | 72.38 [68.50 to 76.30]

13. Secondary Outcome: Change in Family Caregiver Knowledge (as Measured by the Surgery-Related Knowledge Tool)
Description: Mean family caregiver knowledge scores from baseline to 3 months post-discharge were calculated. T-tests were used to assess differences in knowledge between the intervention and control arm at different timepoints.
  Score range: 0-10. Mean: 8.24 with a standard deviation of 1.19. Higher score means better outcome.
Time Frame: Outcomes are measured at baseline, 1 month, and 3 months post-discharge
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Group I (MSM Intervention) | Group II (Attention Control)
Number analyzed (Participants) | 94 | 96
T-score
  Baseline | 8.00 (1.16) | 7.64 (1.42)
  1 month post-discharge: number analyzed (Participants) | 79 | 74
  1 month post-discharge | 8.76 (0.85) | 8.45 (0.91)
  3 months post-discharge: number analyzed (Participants) | 80 | 78
  3 months post-discharge | 8.69 (0.91) | 8.15 (1.26)

14. Secondary Outcome: Change in Patient Knowledge (as Measured by the Surgery-Related Knowledge Tool)
Description: Mean patient knowledge scores from baseline to 3 months post-discharge were calculated. T-tests were used to assess differences in knowledge between the intervention and control arm at different timepoints.
  Score range: 0-10. Mean: 8.42 with a standard deviation of 1.16. Higher score means better outcome.
Time Frame: Outcomes are measured at baseline, 1 month, and 3 months post-discharge
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Group I (MSM Intervention) | Group II (Attention Control)
Number analyzed (Participants) | 94 | 96
T-score
  Baseline | 7.98 (1.25) | 7.98 (1.03)
  1 month post-discharge: number analyzed (Participants) | 81 | 75
  1 month post-discharge | 9.00 (1.18) | 8.48 (1.11)
  3 months post-discharge: number analyzed (Participants) | 93 | 93
  3 months post-discharge | 8.82 (1.00) | 8.50 (0.90)

ADVERSE EVENTS:
Time Frame: This is an intervention trial that lasts 3 months post-treatment with no blood draws, procedures, etc. Since this is not a drug trial, patients and caregivers were not assessed for specific adverse events however, 1 patient died during the study due to acute respiratory failure with hypoxia, not due to study participation. The time frame where each participant was monitored for death was during the 3 months post-discharge.
Description: Since this is not a drug trial, adverse events were not recorded.
Arm/Group | Group I (MSM Intervention) | Group II (Attention Control)
All-Cause Mortality (participants affected / at risk) | 1/188 | 0/192
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-02): https://cdn.clinicaltrials.gov/large-docs/07/NCT03686007/Prot_SAP_000.pdf
  • Informed Consent Form (2023-04-07): https://cdn.clinicaltrials.gov/large-docs/07/NCT03686007/ICF_001.pdf